CLINICAL TRIAL: NCT00622102
Title: Testing Strategies to Improving Warfarin Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Aetna, Inc. (Industry)
Responsible Party: Stephen E. Kimmel, M.D., M.S.C.E., University of Pennsylvania School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 806634
Record Dates: First submitted 2008-01-15; First posted 2008-02-22 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Atrial Fibrillation; Deep Venous Thrombosis; Dilated Cardiomyopathies
Keywords: warfarin; adherence; Mechanical heart valves
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 50% of the consenting subjects will take part in the lottery and use the Med-eMonitor as a device to monitor adherence
  Interventions: Behavioral: Lottery arm (Lottery and Med-eMonitor)
- 2 (Other): 50% of the consenting subjects will use only the Med-eMonitor as a device to monitor adherence
  Interventions: Behavioral: Non-Lottery (Med-eMonitor only)

INTERVENTIONS:
Behavioral: Lottery arm (Lottery and Med-eMonitor) — Lottery and Med-eMonitor
  Arms: 1
Behavioral: Non-Lottery (Med-eMonitor only) — Med-eMonitor only
  Arms: 2

SUMMARY:
We are performing a research study to learn more about the control of an individual's blood thinning (anticoagulation) on warfarin. Individuals from an anticoagulation clinic are being asked to participate in order to see if a lottery which provides the opportunity to win money in combination with the use of the Med-eMonitor might be useful in helping patients to achieve better control of their anticoagulation therapy. Half of the participants will be enrolled in the lottery arm and the other half will be a control group who will receive the Med-eMonitor only.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old age or older
* On warfarin managed at the AC clinic
* Target INR 2.0-3.0 or 2.5-3.5
* At maintenance phase of therapy (defined as stable INR with stable warfarin dosing over at least 2 consecutive visits)

Exclusion Criteria:

* Do not have access to telephone line
* Unwillingness to participate or to sign a consent form(refusal)
* Inability to participate because of advances dementia, advanced Alzheimer's disease or other impairment affecting ability to provide informed consent and/or quality data or utilize the Med-eMonitor
* Participation in a current study that does not permit participation in another study
* End stage or terminal illness with anticipated life expectancy of 6 months or less
* INR over the upper limit for the individual's range at the time of enrollment (e.g.,>3.0 or >3.5, depending on the target range)
* Diagnosed with antiphospholipid antibody syndrome or abnormal INR prior to starting warfarin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
anticoagulation control | six months

SECONDARY OUTCOMES:
adherence | six months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Volpp, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania Anticoagulation Management Center, Philadelphia, Pennsylvania, United States